CLINICAL TRIAL: NCT02320149
Title: A Randomized, Multicenter, Double-blind, Placebocontrolled Study to Evaluate the Efficacy and Safety of 1.5 mg/kg Per Day of Sarecycline Compared to Placebo in the Treatment of Acne Vulgaris
Brief Title: Study to Evaluate Safety & Efficacy of Sarecycline in Treatment of Acne
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SC1401; NCT02651012 (obsolete NCT alias)
Record Dates: First submitted 2014-12-15; First posted 2014-12-19 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Acne Vulgaris
Keywords: acne
MeSH Terms: conditions — Acne Vulgaris | interventions — sarecycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sarecycline (Experimental): Sarecycline tablets, 1.5 milligram(mg)/kilogram(kg)/day, taken orally once daily for 12 weeks.
  Interventions: Drug: Sarecycline
- Placebo (Placebo Comparator): Placebo-matching sarecycline tablets, taken orally once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sarecycline — 1.5 mg/kg/day taken orally at the same time each day,
  Arms: Sarecycline
Drug: Placebo — Placebo-matching sarecycline tablets taken orally at the same time each day.
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of an approximate 1.5mg/kg/day dose of oral sarecycline compared to placebo in the treatment of moderate to severe facial acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent or assent form
* Male/female, 9 to 45 years of age, inclusive
* Body weight between 33 and 136 kg, inclusive
* Facial acne vulgaris with:
* 20-50 inflammatory lesions (papules, pustules and nodules) 30-100 noninflammatory lesions (open and closed comedones)
* No more than 2 nodules
* IGA score of moderate (3) or severe (4)
* Negative urine pregnancy test at baseline - females of childbearing potential
* Agrees to use an effective method of contraception throughout the study
* Refrain from use of any other acne medications and medicated cleansers, and avoid excessive sun exposure and tanning booths for duration of study
* Able to fulfill the requirements of protocol, indicated willingness to participate in the study and agrees to all study procedures (including mandatory photography) by providing written informed consent/assent and an authorization to disclose protected health information (PHI)

Exclusion Criteria:

* Has a dermatological condition of the face that could interfere with the clinical evaluations
* Has a history of any of the following:
* Allergy to tetracycline-class antibiotics or to any ingredient in the study drug
* Pseudomembranous colitis or antibiotic associated colitis
* Treated for any type of cancer within the last 6 months
* Has known resistance to other tetracyclines
* Has received any of the following treatments within 12 weeks of screening:
* Systemic retinoids
* Systemic corticosteroids
* Androgens/anti-androgenic therapy (eg, anabolic steroids, spironolactone)
* Non-medicated procedures for the treatment of acne (eg, laser, light or ThermaClear)
* Has used any acne affecting treatment without an appropriate washout period
* Has initiated hormonal contraceptive use within 12 weeks prior to screening or plans to initiate or switch hormonal contraceptive products during the study period
* Is pregnant, lactating or planning a pregnancy during the study period
* Has any other disorder causing hyperandrogenism including, but not limited to polycystic ovary syndrome, adrenal or ovarian tumors, Cushings disease or congenital adrenal hyperplasia
* Has drug-induced acne
* Has significant intercurrent illness, psychiatric disposition or other factors that, in the opinion of the Investigator or Medical Monitor, precludes participation in the study
* Is currently participating, or has participated within 30 days prior to the screening period in an investigational drug or device study
* Has previously participated in any clinical trial involving the use of sarecycline
* Is judged by the Investigator to be unsuitable for any reason

Ages: 9 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 968 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Kaoukhov, MD, Study Director — Warner Chilcott, an Affiliate of Allergan plc
Locations (57):
- United States (57):
  - Warner Chilcott Research Site (Site #155), Beverly Hills, California
  - Warner Chilcott Research Site (Site #129), Encino, California
  - Warner Chilcott Research Site (Site #150), La Mesa, California
  - Warner Chilcott Research Site (Site #136), Los Angeles, California
  - Warner Chilcott Research Site (Site #147), Sacramento, California
  - Warner Chilcott Research Site (Site #123), San Diego, California
  - Warner Chilcott Research Site (Site #125), San Diego, California
  - Warner Chilcott Research Site (Site #139), Santa Rosa, California
  - Warner Chilcott Research Site (Site #157), Tustin, California
  - Warner Chilcott Research Site (Site #122), Denver, Colorado
  - Warner Chilcott Research Site (Site #148), Wheat Ridge, Colorado
  - Warner Chilcott Research Site (Site #133), New Haven, Connecticut
  - Warner Chilcott Research Site (Site #130), Boca Raton, Florida
  - Warner Chilcott Research Site (Site #152), Boynton Beach, Florida
  - Warner Chilcott Research Site (Site #102), Miami, Florida
  - Warner Chilcott Research Site (Site #145), Miami, Florida
  - Warner Chilcott Research Site (Site #140), North Miami Beach, Florida
  - Warner Chilcott Research Site (Site #151), Orange Park, Florida
  - Warner Chilcott Research Site (Site #108), Sanford, Florida
  - Warner Chilcott Research Site (Site #110), West Palm Beach, Florida
  - Warner Chilcott Research Site (Site #154), Atlanta, Georgia
  - Warner Chilcott Research Site (Site #120), Augusta, Georgia
  - Warner Chilcott Research Site (Site #124), Boise, Idaho
  - Warner Chilcott Research Site (Site #106), Chicago, Illinois
  - Warner Chilcott Research Site (Site #112), Plainfield, Indiana
  - Warner Chilcott Research Site (Site #113), South Bend, Indiana
  - Warner Chilcott Research Site (Site #117), Louisville, Kentucky
  - Warner Chilcott Research Site (Site #135), Lake Charles, Louisiana
  - Warner Chilcott Research Site (Site #153), Metairie, Louisiana
  - Warner Chilcott Research Site (Site #137), Detroit, Michigan
  - Warner Chilcott Research Site (Site #111), Warren, Michigan
  - Warner Chilcott Research Site (Site #119), St Louis, Missouri
  - Warner Chilcott Research Site (Site #138), Omaha, Nebraska
  - Warner Chilcott Research Site (Site #103), Henderson, Nevada
  - Warner Chilcott Research Site (Site #127), Verona, New Jersey
  - Warner Chilcott Research Site (Site #146), New York, New York
  - Warner Chilcott Research Site (Site #132), New York, New York
  - Warner Chilcott Research Site (Site #134), Smithtown, New York
  - Warner Chilcott Research Site (Site #107), High Point, North Carolina
  - Warner Chilcott Research Site (Site #126), Cincinnati, Ohio
  - Warner Chilcott Research Site (Site #143), Warren, Ohio
  - Warner Chilcott Research Site (Site #149), Gresham, Oregon
  - Warner Chilcott Research Site (Site #131), Portland, Oregon
  - Warner Chilcott Research Site (Site #114), Greer, South Carolina
  - Warner Chilcott Research Site (Site #128), Knoxville, Tennessee
  - Warner Chilcott Research Site (Site #109), Nashville, Tennessee
  - Warner Chilcott Research Site (Site #116), Austin, Texas
  - Warner Chilcott Research Site (Site #104), Dallas, Texas
  - Warner Chilcott Research Site (Site #115), El Paso, Texas
  - Warner Chilcott Research Site (Site #142), Houston, Texas
  - Warner Chilcott Research Site (Site #105), Houston, Texas
  - Warner Chilcott Research Site (Site #101), Plano, Texas
  - Warner Chilcott Research Site (Site #118), San Antonio, Texas
  - Warner Chilcott Research Site (Site #156), Layton, Utah
  - Warner Chilcott Research Site (Site #141), Salt Lake City, Utah
  - Warner Chilcott Research Site (Site #121), Charlottesville, Virginia
  - Warner Chilcott Research Site (Site #144), Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Sarecycline: Sarecycline tablets, 1.5 mg/kg/day, taken orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | Sarecycline | Placebo
Started | 483 | 485
Completed | 420 | 405
Not Completed | 63 | 80
Not completed — Adverse Event | 3 | 7
Not completed — Withdrawal of Consent | 28 | 32
Not completed — Lost to Follow-up | 21 | 34
Not completed — Protocol Violation | 2 | 1
Not completed — Noncompliance with Study Treatment | 7 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Other Miscellaneous Reasons | 2 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sarecycline | Placebo | Total
Number analyzed (Participants) | 483 | 485 | 968
Age, Customized [Number; unit: participants]
  ≥9 and <12 Years | 4 | 6 | 10
  ≥12 and <18 Years | 241 | 235 | 476
  ≥18 Years | 238 | 244 | 482
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 268 | 271 | 539
  Male | 215 | 214 | 429
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 377 | 377 | 754
  Black or African American | 80 | 79 | 159
  Asian | 11 | 9 | 20
  American Indian or Alaska Native | 2 | 3 | 5
  Native Hawaiian or other Pacific Islander | 2 | 3 | 5
  Multiple races | 11 | 14 | 25
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 144 | 143 | 287
  Not Hispanic or Latino | 339 | 342 | 681
Inflammatory Lesion Counts [Mean (Standard Deviation); unit: lesion count] — Facial area lesion counts were made at forehead, left and right cheeks, nose, and chin. Inflammatory lesion counts were defined as: papule: a solid, elevated lesion <0.5 cm in diameter with surrounding erythematous halo; pustule: an elevated lesion containing pus <0.5 cm in diameter with surrounding erythematous halo; nodule: palpable solid erythematous lesion >0.5 cm in diameter; has depth, not necessarily elevated.
  lesion count | 29.7 (8.7) | 30.2 (9.6) | 30.0 (9.2)
Investigator's Global Assessment (IGA) Score - Face [Mean (Standard Deviation); unit: score on a scale] — The investigator assessed the participant's inflammatory lesions on the face using the IGA 5-point scale. The scale ranges from 0 (best): clear, no evidence of papules or pustules to 4 (worst): severe, inflammatory lesions are more apparent, many papules/pustules, there may or may not be a few nodulocytic lesions.
  score on a scale | 3.1 (0.4) | 3.2 (0.4) | 3.1 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Facial Inflammatory Lesion Counts at Week 12
Description: Facial area lesion counts were made at the forehead, left and right cheeks, nose, and chin at baseline and at each treatment period visit. Inflammatory lesion counts were based on the following definitions: papule: a solid, elevated lesion < 0.5 centimeter (cm) in diameter (by inspection) with surrounding erythematous halo; pustule: an elevated lesion containing pus < 0.5 cm in diameter (by inspection) with surrounding erythematous halo; nodule: palpable solid erythematous lesion > 0.5 cm in diameter (by inspection); has depth, not necessarily elevated. A negative change from Baseline indicates that the number of inflammatory lesions decreased. Analyses were based on Analysis of Covariance (ANCOVA) model for the endpoint with treatment group and pooled study center as factors and baseline value as a covariate.
Time Frame: Baseline (Day 1) to Week 12
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
lesion count | -15.3 (0.6) | -10.1 (0.6)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — Analyses were based on ANCOVA model for the endpoint with treatment group and pooled study center as factors and baseline value as a covariate; Least Squares Mean Difference = -5.2, 95% CI 2-sided [-6.7 to -3.6] — sarecycline - placebo

2. Primary Outcome: Percentage of Participants With Investigator Global Assement (IGA) Success at Week 12
Description: The investigator assessed the participant's inflammatory lesions on the face using the IGA 5-point scale. The scale ranges from 0 (best): clear, no evidence of papules or pustules to 4 (worst): severe, inflammatory lesions are more apparent, many papules/pustules, there may or may not be a few nodulocytic lesions. Success was defined as at least a 2-point decrease (improvement) from Baseline on the IGA assessment as well as a score of clear (0) or almost clear (1). The percentage of participants who achieved success is reported.
Time Frame: Baseline (Day 1) to Week 12
Population: ITT population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
percentage of participants | 21.9 | 10.5
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-values were based on the test of general association between the response and treatment group using Cochran-Mantel-Haenszel test with pooled site as stratification factor; Treatment Rate Difference = 11.05, 95% CI 2-sided [6.39 to 15.72] — sarecycline - placebo

3. Secondary Outcome: Percent Change From Baseline in Facial Inflammatory Lesion Counts at Week 12
Description: Facial area lesion counts were made at the forehead, left and right cheeks, nose, and chin at baseline and at each treatment period visit. Inflammatory lesion counts were based on the following definitions: papule: a solid, elevated lesion < 0.5 centimeter (cm) in diameter (by inspection) with surrounding erythematous halo; pustule: an elevated lesion containing pus < 0.5 cm in diameter (by inspection) with surrounding erythematous halo; nodule: palpable solid erythematous lesion > 0.5 cm in diameter (by inspection); has depth, not necessarily elevated. A negative change from Baseline indicates that the number of inflammatory lesions decreased. Analyses were based on ANCOVA model for the endpoint with treatment group and pooled study center as factors and baseline value as a covariate.
Time Frame: Baseline (Day 1) to Week 12
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percent change in lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
percent change in lesion count | -51.8 (1.9) | -35.1 (2.0)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Percent Change from Baseline to Week 12; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -16.7, 95% CI 2-sided [-21.9 to -11.6] — sarecycline - placebo

4. Secondary Outcome: Percent Change From Baseline in Facial Inflammatory Lesion Counts at Week 9
Description: as for outcome 3
Time Frame: Baseline (Day 1) to Week 9
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percent change in lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
percent change in lesion count | -47.4 (1.7) | -34.9 (1.7)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Percent Change from Baseline to Week 9; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -12.5, 95% CI [-16.9 to -8.0] — sarecycline - placebo

5. Secondary Outcome: Percent Change From Baseline in Facial Inflammatory Lesion Counts at Week 6
Description: as for outcome 3
Time Frame: Baseline (Day 1) to Week 6
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percent change in lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
percent change in lesion count | -42.2 (1.6) | -28.9 (1.6)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Percent Change from Baseline to Week 6; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -13.3, 95% CI 2-sided [-17.5 to -9.1] — sarecycline - placebo

6. Secondary Outcome: Percent Change From Baseline in Facial Inflammatory Lesion Counts at Week 3
Description: as for outcome 3
Time Frame: Baseline (Day 1) to Week 3
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percent change in lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
percent change in lesion count | -29.6 (1.5) | -22.4 (1.5)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Percent Change from Baseline to Week 3; Test type: Superiority; p = 0.0003, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -7.2, 95% CI 2-sided [-11.1 to -3.3] — sarecycline - placebo

7. Secondary Outcome: Absolute Change From Baseline in Facial Inflammatory Lesion Counts at Week 9
Description: Facial area lesion counts were made at the forehead, left and right cheeks, nose, and chin at baseline and at each treatment period visit. Inflammatory lesion counts were based on the following definitions: papule: a solid, elevated lesion < 0.5 cm in diameter (by inspection) with surrounding erythematous halo; pustule: an elevated lesion containing pus < 0.5 cm in diameter (by inspection) with surrounding erythematous halo; nodule: palpable solid erythematous lesion > 0.5 cm in diameter (by inspection); has depth, not necessarily elevated. A negative change from Baseline indicates that the number of inflammatory lesions decreased. Analyses were based on ANCOVA model for the endpoint with treatment group and pooled study center as factors and baseline value as a covariate.
Time Frame: Baseline (Day 1) to Week 9
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
lesion count | -13.9 (0.5) | -10.0 (0.5)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Change from Baseline to Week 9; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -3.9, 95% CI 2-sided [-5.3 to -2.5] — sarecycline - placebo

8. Secondary Outcome: Absolute Change From Baseline in Facial Inflammatory Lesion Counts at Week 6
Description: as for outcome 7
Time Frame: Baseline (Day 1) to Weeks 6
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
lesion count | -12.5 (0.5) | -8.4 (0.5)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Change from Baseline to Week 6; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -4.1, 95% CI 2-sided [-5.4 to -2.9] — sarecycline - placebo

9. Secondary Outcome: Absolute Change From Baseline in Facial Inflammatory Lesion Counts at Week 3
Description: as for outcome 7
Time Frame: Baseline (Day 1) to Week 3
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
lesion count | -8.5 (0.4) | -6.4 (0.4)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Change from Baseline to Week 3; Test type: Superiority; p = 0.0005, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -2.1, 95% CI 2-sided [-3.3 to -0.9] — sarecycline - placebo

10. Secondary Outcome: Percent Change From Baseline in Facial Noninflammatory Lesion Counts at Week 12
Description: Facial area lesion counts were made at the forehead, left and right cheeks, nose, and chin at baseline and at each treatment period visit. Noninflammatory lesion counts were based on the following definitions: open comedones (blackheads): noninfected plugged hair follicle with a dilated/open orifice, black in color; closed comedones (whiteheads): noninfected plugged hair follicle with a small (microscopic) opening at the surface of the skin. A negative change from Baseline indicates that the number of noninflammatory lesions decreased. Analyses were based on ANCOVA model for the endpoint with treatment group and pooled study center as factors and baseline value as a covariate.
Time Frame: Baseline (Day 1) to Week 12
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percent change in lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
percent change in lesion count | -27.0 (5.6) | -22.7 (5.6)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Percent Change from Baseline to Week 12; Test type: Superiority; p = 0.5786, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -4.3, 95% CI 2-sided [-19.4 to 10.8] — sarecycline - placebo

11. Secondary Outcome: Percent Change From Baseline in Facial Noninflammatory Lesion Counts at Week 9
Description: as for outcome 10
Time Frame: Baseline (Day 1) to Week 9
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percent change in lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
percent change in lesion count | -20.8 (5.3) | -18.0 (5.3)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Percent Change from Baseline to Week 9; Test type: Superiority; p = 0.6969, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -2.8, 95% CI 2-sided [-17.1 to 11.4] — sarecycline - placebo

12. Secondary Outcome: Percent Change From Baseline in Facial Noninflammatory Lesion Counts at Week 6
Description: as for outcome 10
Time Frame: Baseline (Day 1) to Week 6
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percent change in lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
percent change in lesion count | -14.6 (6.6) | -17.6 (6.6)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Percent Change from Baseline to Week 6; Test type: Superiority; p = 0.7377, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 3.0, 95% CI 2-sided [-14.7 to 20.7] — sarecycline - placebo

13. Secondary Outcome: Percent Change From Baseline in Facial Noninflammatory Lesion Counts at Week 3
Description: as for outcome 10
Time Frame: Baseline (Day 1) to Week 3
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percent change in lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
percent change in lesion count | -8.0 (4.4) | -14.3 (4.3)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Percent Change from Baseline to Week 3; Test type: Superiority; p = 0.2861, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = 6.4, 95% CI 2-sided [-5.3 to 18.1] — sarecycline - placebo

14. Secondary Outcome: Absolute Change From Baseline in Facial Noninflammatory Lesion Counts at Week 12
Description: as for outcome 10
Time Frame: Baseline (Day 1) to Week 12
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
lesion count | -15.1 (0.9) | -11.2 (0.9)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Change from Baseline to Week 12; Test type: Superiority; p = 0.0014, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -3.9, 95% CI 2-sided [-6.3 to -1.5] — sarecycline - placebo

15. Secondary Outcome: Absolute Change From Baseline in Facial Noninflammatory Lesion Counts at Week 9
Description: as for outcome 10
Time Frame: Baseline (Day 1) to Week 9
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
lesion count | -13.0 (0.8) | -9.6 (0.8)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Change from Baseline to Week 9; Test type: Superiority; p = 0.0010, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -3.4, 95% CI 2-sided [-5.5 to -1.4] — sarecycline - placebo

16. Secondary Outcome: Absolute Change From Baseline in Facial Noninflammatory Lesion Counts at Week 6
Description: as for outcome 10
Time Frame: Baseline (Day 1) to Week 6
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
lesion count | -10.6 (0.7) | -8.6 (0.7)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Change from Baseline to Week 6; Test type: Superiority; p = 0.0371, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-4.0 to -0.1] — sarecycline - placebo

17. Secondary Outcome: Absolute Change From Baseline in Facial Noninflammatory Lesion Counts at Week 3
Description: as for outcome 10
Time Frame: Baseline (Day 1) to Week 3
Population: ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: lesion count
Arm/Group | Sarecycline | Placebo
Number analyzed (Participants) | 483 | 485
lesion count | -7.9 (0.6) | -7.1 (0.6)
Statistical Analysis 1: Comparison: Sarecycline vs Placebo; Change from Baseline to Week 3; Test type: Superiority; p = 0.3806, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.8, 95% CI 2-sided [-2.5 to 1.0] — sarecycline - placebo

ADVERSE EVENTS:
Time Frame: Up to 20.7 Weeks
Description: The number of participants at risk for Serious Adverse Events and Adverse Events were based on the Safety Population that included all participants who received at least one dose of study treatment. Two participants in the sarecycline arm and two in the placebo arm did not receive study treatment.
Arm/Group | Sarecycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/481 | 0/483
Serious Adverse Events (participants affected / at risk) | 3/481 | 5/483
Other Adverse Events (participants affected / at risk) | 0/481 | 0/483
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sarecycline (N=481) | Placebo (N=483)
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Suicide attempt (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Miscarriage of partner (Social circumstances) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2015-12-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT02320149/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT02320149/SAP_001.pdf